CLINICAL TRIAL: NCT01031212
Title: A Phase I Study of ASA 404 in Combination With Carboplatin/Paclitaxel/Cetuximab in Patients With Refractory Solid Tumors
Brief Title: ASA404 in Combination With Carboplatin/Paclitaxel/Cetuximab in Treating Patients With Refractory Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The investigator has left the institution (UCSF) prior to study start-up
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sarita Dubey, MD, University of California, San Franciso
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF-09997; H53469-35218 (Other: UCSF Committee on Human Research)
Record Dates: First submitted 2009-12-08; First posted 2009-12-14 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Tumors
Keywords: cancer; neoplasms; adult solid tumor; antineoplastic agents
MeSH Terms: conditions — Neoplasms | interventions — vadimezan; Cetuximab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ASA404 — Administered intravenously over 20 minutes weekly after chemotherapy
  Other Names: 5-6-dimethylxanthenone-4-acetic acid; DMXAA; AS1404
Drug: Cetuximab — Administered at 400mg/m2 over 120 minutes on day -7 and then 250mg/m2 over 60 minutes weekly thereafter
  Other Names: Erbitux
Drug: Carboplatin — Administered at fixed dose of AUC 6 intravenously on day 1 of each 3-week cycle
  Other Names: Paraplatin
Drug: Paclitaxel — Administered over 3 hours at a fixed dose of 175mg/m2 intravenously on day 1 of each 3-week cycle
  Other Names: Taxol

SUMMARY:
This phase I trial is studying the side effects and best dose of an investigational drug called DMXAA (5-6-dimethylxanthenone-4-acetic acid) or ASA404 when given together with carboplatin, paclitaxel and cetuximab to treat patients with refractory solid tumors.

DETAILED DESCRIPTION:
Phase I 3+3 dose escalation design in patients with solid tumors who have been previously treated with chemotherapy or for whom no standard treatment options exist. Carboplatin, paclitaxel and cetuximab will be administered in standard doses. The dose of ASA404 will be escalated under predefined levels. One treatment cycle constitutes 3 weeks. A minimum of 3 patients will be entered at each treatment level, to be expanded to 6 subjects if dose limiting toxicities (DLT) are observed. If no more than one in six patients has DLT, additional patients will be enrolled at a higher dose. Once a maximum tolerated dose (MTD) has been established, the tolerability of this dose will be tested in a total of 12 patients. The anticipated sample size is 18-24 patients.

Carboplatin and paclitaxel are chosen as the chemotherapy back bone since they are commonly used in combination in multiple tumors. Cetuximab has been chosen as the EGFR inhibitor because the combination of platinum based therapy with cetuximab is effective in lung and head and neck cancers. In addition the safety and activity of carboplatin/paclitaxel with ASA 404 has already been demonstrated. A weekly schedule of ASA is chosen because 1) the safety of the weekly schedule has been tested 2) preclinical studies confirm enhanced activity with frequent administration 3) provides an opportunity to evaluate the safety and pharmacokinetics of ASA 404 with weekly cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed malignancy of advanced, incurable solid tumor
* Progression following standard therapy, or no acceptable standard treatment options, or eligible if standard therapy consists of a platinum-based doublet
* Measurable or evaluable disease. Measurable disease required for enrollment in dose expansion cohort at MTD
* ECOG 0-2
* Baseline neuropathy grade ≤ 1
* leukocytes >3,000/mcL
* absolute neutrophil count >1,500/mcL
* platelets >100,000/mcL
* total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) <1.5 X institutional ULN
* creatinine within 1.5 x normal institutional limits OR creatinine clearance >60 mL/min/1.73 m2
* Ability to give written informed consent and willingness to comply with requirements of the protocol
* Women of child-bearing potential must have a negative pregnancy test within 14 days of beginning study drug and agree to use an effective method of birth control during treatment and for six months after last dose of study drug
* Male patients whose sexual partners are women of reproductive potential must be surgically sterile or agree to use a double method of contraception during the study and for six months after last dose of study drug. One of method must be a condom
* Patients with known brain metastases should have "stable disease" defined as no growth over a 6 week period after definitive therapy (surgical or RT), and off steroids and anticonvulsive therapy

Exclusion Criteria:

* Chemotherapy, hormonal therapy or biologic therapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to the start of study therapy or not recovered to < grade 2 from adverse events due to prior agents
* Prior therapy with EGFR inhibitors is permitted
* Patients receiving palliative radiation therapy <2 weeks earlier. Patients must have recovered from all toxicities of radiation
* Receiving any other investigational agents
* Any severe and/or uncontrolled intercurrent medical conditions or other conditions that could affect participation in the study
* Any of the following cardiac abnormalities: unstable angina pectoris, including Prinzmetal variant angina, New York Heart Association (NYHA) Classification for Congestive Heart Failure Grade III or greater, myocardial infarction or stroke ≤ 12 months prior to study treatment, long QT syndrome, baseline 12 lead ECG QTc of >450msec per central evaluation, history of sustained ventricular tachycardia, history of ventricular fibrillation or Torsades de Pointes, right bundle branch block and left anterior hemiblock (bifascicular block), bradycardia (<50 beats per minute)
* Concomitant use of drugs with a risk of causing Torsades de Pointes
* PT/PTT > 1.5 x ULN
* Receiving full-dose anticoagulation (low-dose warfarin for a central line allowed)
* History of another primary malignancy less than 5 years prior, except non-melanoma skin cancer or cervical cancer in-situ
* Major surgery ≤ 4 weeks prior (requiring general anesthesia or respiratory assistance)(endoscopic exams with diagnostic intent allowed)
* Minor surgery ≤ 2 weeks prior (not requiring general anesthesia or respiratory assistance)
* Insertion of vascular access device allowed
* Not recovered from surgery-related complications
* Systolic BP >160mmHg and/or diastolic BP >90mmHg while on medication for hypertension
* Hemoptysis associated with chest malignancy <4 weeks (>1 teaspoon)
* History of hypersensitivity reactions to TAXOL or other drugs formulated in Cremophor® EL (polyoxyethylated castor oil)
* History of severe allergic reactions to cisplatin or other platinum-containing compounds
* History of acute hemorrhagic events requiring hospital admission or blood transfusion
* Pregnant or lactating women
* Fertile women and men not willing to comply with birth control instructions
* Any condition that compromises compliance with objectives and procedures of this protocol, as judged by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | During cycle 1 (4 weeks)

SECONDARY OUTCOMES:
The number and percentage of subjects experiencing one or more AEs will be summarized by dose cohort, relationship to study drug, and severity | Within 30 days after study treatment, or until resolution of AE
Pharmacokinetics of ASA404 in combination with other agents | 48 hours after cycle 1, day 1
Disease response by RECIST criteria | until progression
Assess biological correlates of antitumor activity by measuring serum 5HIAA, VEGF, bFGF, PLGF, sVEGFR2, FGF 23, serum apoptotic markers (M30/M65) | 4 weeks after treatment end
DNA analysis of FGFR1 and VEGF polymorphism | 4 weeks after treatment ends

CONTACTS AND LOCATIONS:
Overall Officials: Sarita Dubey, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States